CLINICAL TRIAL: NCT03494270
Title: A Randomized, Open, Parallel, Multicenter, Phase 4 Study to Compare High-intensity Rosuvastatin to Moderate-intensity Rosuvastatin/Ezetimibe in Atherosclerotic Cardiovascular Disease (ASCVD) Patients
Brief Title: High-intensity Rosuvastatin and Moderate-intensity Rosuvastatin/Ezetimibe in ASCVD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC033
Record Dates: First submitted 2018-04-02; First posted 2018-04-11 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: ASCVD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvamibe Tab (Experimental): Rosuvastatin 10mg/Ezetimibe 10mg qd for 24 weeks
  Interventions: Drug: Rosuvamibe
- Monorova Tab (Active Comparator): Rosuvastatin 20mg qd for 24 weeks
  Interventions: Drug: Monorova

INTERVENTIONS:
Drug: Rosuvamibe — Rosuvastatin 10mg/Ezetimibe 10mg
  Arms: Rosuvamibe Tab
Drug: Monorova — Rosuvastatin 20mg
  Arms: Monorova Tab

SUMMARY:
This study will evaluate the efficacy and safety of high-intensity rosuvastatin and moderate-intensity rosuvastatin/ezetimibe in ASCVD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 to 75 years
2. Patients diagnosed with ASCVD (coronary artery disease)

   * acute coronary syndrome
   * history of myocardial infarction (MI)
   * stable or unstable angina
   * history of coronary revascularization
   * stroke or transient ischemic attack (TIA)
   * peripheral arterial disease, history of peripheral arterial revascularization
3. Taking a stable dose of a statin or a lipid-lowering agent of ezetimibe over 4 weeks before randomization
4. Written informed consent

Exclusion Criteria:

1. Administration of other lipid lowering agents than statin or ezetimibe within 3 months prior to screening visit
2. Fasting triglyceride ≥ 400 mg/dL
3. History of muscular disease or rhabdomyolysis due to use of statin
4. Hypersensitive to rosuvastatin or ezetemibe
5. Contraindications stated in the SPC of rosuvastatin or rosuvastatin/ezetimibe including the following:

   ① Severe renal disease (CrCL < 30mL/min: Cockcroft-gault formula or estimated GFR (MDRD) < 30mL/min/1.73m2)

   ② ALT, AST > 3x ULN or history of active liver disease

   ③ CPK > 3x ULN
6. Administration of other investigational products within 30 days prior to screening visit
7. Other than the above who is deemed to be ineligible to participate in the trial by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 in LDL-C level | Baseline, Week 12

SECONDARY OUTCOMES:
Change from baseline to week 12 and week 24 in total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), triglycerides (TG), Non-HDL cholesterol, Apolipoprotein A1, and Apolipoprotein B | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in high-sensitivity C-reactive protein (hs-CRP) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in fasting plasma glucose (FPG) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in homeostasis model assessment for insulin resistance (HOMA-IR) | Baseline, Week 12, Week 24
Proportion of subjects achieving LDL-C < 70mg/dL | Baseline, Week 12, Week 24
Occurrence of Statin-Associated Muscle Symptoms (SAMS) | Up to 24 weeks
Proportion of subjects with CPK 4 x upper limit of normal (ULN) or 10 x ULN | Baseline, Week 12, Week 24
Proportion of subjects with AST or ALT levels elevated to 4 x ULN or 10 x ULN | Baseline, Week 12, Week 24
Occurrence of MACCE (Major Adverse Cardiovascular and Cerebrovascular Event) | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi H, Kang SH, Jeong SW, Yoon CH, Youn TJ, Song WH, Jeon DW, Lim SW, Lee JH, Cho SW, Chae IH, Kim CH. Lipid-Lowering Efficacy of Combination Therapy With Moderate-Intensity Statin and Ezetimibe Versus High-Intensity Statin Monotherapy: A Randomized, Open-Label, Non-Inferiority Trial From Korea. J Lipid Atheroscler. 2023 Sep;12(3):277-289. doi: 10.12997/jla.2023.12.3.277. Epub 2023 Aug 3. PMID 37800112